| Cover page |
|---|
| Title: Individual Follow-up after Rectal Cancer - Focus on the Needs of the Patient (FURCA) |
| [NCT-number not assigned yet] |
| Date: 07 February 2016 |

## Statistical analysis plan for the FURCA-trial

Outcomes will be analyzed using methods for repeated measurements and survival analysis. Any difference between the two groups will be significance tested, and adjusted for covariates, using multiple regression analysis.

Differences in demographics between the two groups will be calculated and significance tested using a chi2-test (dichotomous and categorical data) and t-test (numerical data).

Quality-adjusted life years will be calculated using standard health economic methods and in collaboration with an expert in health economics.

A more detailed plan for statistical analyses will be uploaded.